CLINICAL TRIAL: NCT00008229
Title: A Phase III Multicenter, Randomized, Open-Label Trial Evaluating High Dose Melphalan Plus Holmium-166-DOTMP Versus High Dose Melphalan Alone When Given In Conjuction With Peripheral Blood Stem Cell Transplantation In Patients With Multiple Myeloma
Brief Title: Melphalan With or Without Holmium Ho 166 DOTMP Followed by Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1542.00; FHCRC-1542.00; NEORX-9902; UCLA-0006110; NCI-G00-1892; CDR0000068389 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-01-06; First posted 2004-05-24 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Melphalan; Peripheral Blood Stem Cell Transplantation; holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan
Procedure: peripheral blood stem cell transplantation
Radiation: holmium Ho 166 DOTMP

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radioactive drugs such as holmium Ho 166 DOTMP can kill cancer cells without harming healthy cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of melphalan with or without holmium Ho 166 DOTMP followed by peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of melphalan with or without holmium Ho 166 DOTMP followed by autologous peripheral blood stem cell transplantation in patients with multiple myeloma. II. Compare the response rate and overall survival of these patients treated with these regimens. III. Compare the hematologic recovery rate and time to granulocyte engraftment of these patients treated with these regimens. IV. Compare the toxicity of these regimens in this patient population.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to their beta 2 microglobulin (B2M) test at initial diagnosis (B2M no greater than 4 mg/L vs B2M greater than 4 mg/L vs unknown B2M). Patients are randomized to one of two treatment arms. Prior to stratification and randomization, patients receive a diagnostic dose of holmium Ho 166 DOTMP within days -31 to -10. Patients with adequate skeletal uptake of the diagnostic dose are randomized for therapy. Arm I: Patients receive holmium Ho 166 DOTMP IV over no more than 10 minutes within days -10 to -7 (at least 1 week and no more than 3 weeks after the diagnostic dose), melphalan IV over 20-30 minutes within days -3 to -1 (at least 24 hours prior to autologous peripheral blood stem cell (PBSC) transplantation), and autologous PBSC transplantation on day 0. Arm II: Patients receive melphalan and autologous PBSC transplantation as in arm I. Following transplantation, patients receive filgrastim (G-CSF) daily until blood counts recover. Patients are followed at 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 300 patients (150 per treatment arm) will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed multiple myeloma (diagnosis within 12 months of study) and scheduled to undergo autologous peripheral blood stem cell transplantation Prior diagnosis of monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SMM) allowed if the criteria for diagnosis of multiple myeloma was met within 12 months of study Serum or urinary M-protein confirmation of diagnosis (IgA, IgD, IgG, IgE, or light chain proteins) At least 10% plasma cells in bone marrow Must have received induction therapy without disease progression or relapse after initial response Prior induction therapy must have been completed no more than 6 months before stem cell collection and no more than 9 months before transplantation Must have undergone stem cell mobilization with cyclophosphamide IV and filgrastim (G-CSF) The following diagnoses are excluded: Non-secretory multiple myeloma IgM myeloma Solitary bone or extramedullary plasmacytoma Symptomatic MGUS or SMM Symptomatic indolent multiple myeloma

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2 mg/dL SGPT no greater than 2 times upper limit of normal No clinical evidence of amyloidosis involving the liver Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 30 mL/min No clinical evidence of amyloidosis involving the kidney Cardiovascular: LVEF at least 50% No evidence of amyloidosis on echocardiogram No uncontrolled arrhythmia No symptomatic cardiac disease Pulmonary: FEV1 at least 60% OR FVC at least 60% OR DLCO at least 60% No symptomatic pulmonary disease No clinical evidence of amyloidosis involving the lungs Other: HIV negative No cord compression No other concurrent illness that would preclude survival No clinical evidence of amyloidosis involving the autonomic nervous system or gastrointestinal tract No known allergy to vitamin C Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior thalidomide for myeloma No prior peripheral blood stem cell or bone marrow transplantation No concurrent thalidomide No concurrent interferon Chemotherapy: See Disease Characteristics No prior clarithromycin for myeloma No more than 2 courses of prior induction therapy containing an alkylating agent Endocrine therapy: No concurrent dexamethasone Radiotherapy: No prior radiotherapy to more than 20% of bone marrow No greater than 30 Gy to the spinal cord Surgery: Not specified Other: At least 28 days since prior bisphosphonates No prior new or experimental agents for myeloma No concurrent experimental therapies No concurrent bisphosphonates

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States